CLINICAL TRIAL: NCT04023500
Title: Supporting Oral Self-care of Patients With Periodontitis Through Brief Motivational Interview
Brief Title: Supporting Oral Self-care of Patients With Periodontitis Through Motivational Interview
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Mirkka Järvinen, Principal investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: University of Turku
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Periodontal Diseases; Patient Education; Self-Care
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded, patients and dentist who performs baseline and follow-up measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview (Active Comparator): The MI-intervention is used as a part of normal dental hygienist appointment. Dental hygienists are trained to focus on patients view of their oral health, self-care skills and need for oral-health related behaviour change. They are supposed to use open-ended questions, reflective listening and reinforcing with patients. Dental hygienist support patients in decision making although patients were addressed as an active agent.
  Interventions: Behavioral: Motivational interview vs. prevailing education
- Prevailing education (Active Comparator): In control group prevailing, more professional-centered education is used. Dental hygienist define patients educational needs and give direct instructions how to change behaviour and self-care.
  Interventions: Behavioral: Motivational interview vs. prevailing education

INTERVENTIONS:
Behavioral: Motivational interview vs. prevailing education — In intervention group dental hygienists are trained to focus on patients view of their oral health, self-care skills and need for oral-health related behaviour change. They are supposed to use open-ended questions, reflective listening and reinforcing with patients.
  In control croup dental hygienist defined patients educational needs and gave direct instructions how to change behaviour and self-care.

SUMMARY:
The aim of this study was to evaluate the potential additive effect of Motivational Interviewing (MI) on gingival health and self-care. Our hypothesis was that the Motivational Interviewing would result in improved gingival health and self-care compared to prevailing patient education.

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blinded, controlled clinical trial of 6-month duration involving patients with diagnosed periodontitis. The subjects are randomized to intervention or control group using the randomizing list.

For both groups, necessary non-surgical periodontal treatments will be done. In the intervention group The MI-intervention is used as a part of normal dental hygienist appointment and if patient need more than one visit, MI was used in every visit.

In control group prevailing, more professional-centered education is used. Dental hygienist define patients educational needs and give direct instructions how to change behaviour and self-care.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over 18-year-old
* CPI (Community periodontal index) 3 in at least two sextants and
* Diagnosed parodontitis
* The previous treatment period should have been more than one year ago.

Exclusion Criteria:

* pregnancy (or the planning of pregnancy)
* immunosuppressive illness or a medication,
* hepatitis, HIV, MRSA (methicillin-resistant Staphylococcus aureus)
* a bleeding illness or a anticoagulant (excluding primalan 100-200 mg / a day)
* the labile diabetes
* cytotoxic treatment
* a need for the antibiotic prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BoP) | Up to 6 month
  Change in BoP is measured three times during the study. In the baseline and in the tree- and six-months follow-up.
  Bop is recorded60 seconds after the pocket probing and assessed as present (1) or absent (0) on four surfaces.
Pocket probing depth (PD) | Up to 6 month
  Change in PD is measured three times during the study. In the baseline and in the tree- and six-months follow-up. PD is measured at mesial, distal, lingual and buccal surfaces.
Clinical Attachment Level (CAL) | Up to 6 month
  Change in CAL is measured three times during the study. In the baseline and in the tree- and six-months follow-up. CAL is measured if cemento-enamel junction is uncovered or if there is 6 mm deep or deeper gingival pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Mirkka Järvinen, MNS, Principal Investigator — University of Turku

IPD SHARING:
Plan to Share IPD: No